CLINICAL TRIAL: NCT05465681
Title: A Phase I Clinical Study of Safety and Pharmacokinetics of Single-dose HR20013 for Injection Combined With Dexamethasone in Patients With Malignant Solid Tumors Receiving Cisplatin-based Chemotherapy
Brief Title: Study of HR20013 for Injection in Patients With Malignant Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Fujian Shengdi Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: HR20013-102
Record Dates: First submitted 2022-07-15; First posted 2022-07-20 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2022-06

CONDITIONS: Prevention of Nausea and Vomiting Caused by Highly Emetogenic Chemotherapy

STUDY DESIGN:
Intervention Model Description: HR20013 for injection combined with dexamethasone
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HR20013 for injection+dexamethasone (Experimental)
  Interventions: Drug: HR20013 for injection；dexamethason

INTERVENTIONS:
Drug: HR20013 for injection；dexamethason — HR20013 for injection；Drug for preventing nausea and vomiting caused by chemotherapy.
  dexamethasone: Drug for preventing nausea and vomiting caused by chemotherapy

SUMMARY:
To evaluate the safety and pharmacokinetics of single-dose HR20013 for injection combined with dexamethasone in patients with malignant solid tumors receiving cisplatin-based chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or older, of either gender
2. Has a diagnosed malignant tumor
3. has never been treated with cisplatin and is to receive the first course of cisplatin-based chemotherapy (≥60 mg/m2)
4. Predicted life expectancy of ≥ 3 months
5. Has a performance status (ECOG scale) of 0 to 1
6. Adequate bone marrow, kidney, and liver function
7. Women of childbearing potential must have negative pregnancy test (serum test) results within 72 hours prior to enrollment
8. Able and willing to provide a written informed consent

Exclusion Criteria:

1. Scheduled to receive any radiation therapy to the abdomen or pelvis from Day -7 through Day 8
2. Scheduled to receive any other chemotherapeutic agent with an high emetogenicity level from Day 2 through Day 8
3. Has taken the following agents within the last 48 hours 5-HT3 antagonists, Phenothiazines, Benzamides, Domperidone, Cannabinoids, Benzodiazepines
4. Subjects receiving palonosetron hydrochloride within 14 days before enrollment
5. Subjects who previously received NK-1 receptor antagonists within 14 days prior to enrollment
6. Subjects with a history of myocardial infarction or unstable angina pectoris
7. Subjects with atrioventricular block or cardiac insufficiency
8. Subjects with poor blood pressure control after medication
9. Subjects with symptomatic brain metastases or any symptoms suggestive of brain metastasis or intracranial hypertension
10. Subjects who have experienced emetic events (vomiting or dry vomiting) or nausea within 24 hours prior to the start of cisplatin
11. Participated in clinical trials of other drugs (received experimental drugs)
12. The investigators determined that other conditions were inappropriate for participation in this clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2022-08-30 (Actual); Primary Completion 2023-01-13 (Actual); Study Completion 2023-01-13 (Actual)

PRIMARY OUTCOMES:
AUC0-t ：area under the plasma concentration-time curve from time 0 to the time of the last quantifiable concentration | 0 to 504 hours
AUC0-∞：Area Under the Plasma Concentration-time Curve From Time 0 to Infinity | 0 to 504 hours
Cmax：observed maximum plasma concentration | 0 to 504 hours
Tmax：observed time to reach Cmax | 0 to 504 hours
T1/2z：apparent terminal half-life | 0 to 504 hours

SECONDARY OUTCOMES:
The number of participants with injection site reaction and treatment-related adverse events as assessed by CTCAE v5.0 | 0 to 504 hours
  The number of participants with injection site reaction and treatment-related adverse events as assessed by CTCAE v5.0
Complete response | During the Acute Phase [0-24 hours after the start of cisplatin administration], the Delayed (>24-120 hours) phase, the overall (0-120 hours) phase, >120-168 hours and 0-168 hours
No significant nausea (maximum nausea on a visual analogue scale<25 mm) | During the Acute Phase, the Delayed phase, the overall phase, >120-168 hours and 0-168 hours
No nausea (maximum nausea on a visual analogue scale<5 mm) | During the Acute Phase, the Delayed phase, the overall phase, >120-168 hours and 0-168 hours
No emetic | During the Acute Phase, the Delayed phase, the overall phase, >120-168 hours and 0-168 hours
No rescue medication | During the Acute Phase, the Delayed phase, the overall phase, >120-168 hours and 0-168 hours
Time to treatment failure | During 0-168 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Zhao Y, Ma Y, Yin T, Qin Z, Liu L, Kong G, Zhang R, Huang Y, Zhang L, Zhao H. Pharmacokinetics, safety, and efficacy of mixed formulation of fosrolapitant and palonosetron (HR20013) in combination with dexamethasone in patients with solid tumors scheduled for highly emetogenic cisplatin-based chemotherapy: a phase I trial. BMC Med. 2025 Aug 27;23(1):501. doi: 10.1186/s12916-025-04314-5. PMID 40866861